CLINICAL TRIAL: NCT01342172
Title: Multi-Center Phase Ib/II Trial of Gemcitabine, Cisplatin, Plus Lenalidomide as First-line Therapy for Patients With Metastatic Urothelial Carcinoma
Brief Title: Gemcitabine, Cisplatin, Plus Lenalidomide as First-line Therapy for Patients With Metastatic Urothelial Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Matthew Galsky, Principal Investigator, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 10-1339; NCT01441050 (obsolete NCT alias)
Record Dates: First submitted 2011-04-21; First posted 2011-04-27 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Bladder Cancer; Urothelial Cancer; Chemotherapy; First-line; Metastatic
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasm Metastasis | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): capsules for oral administration
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Patients will receive gemcitabine 1000 mg/m2 IV on days 1 + 8 and cisplatin 70 mg/m2 IV on day 1 of each 21 day cycle. Lenalidomide will be given orally on days 1-14 and the dose will be escalated in successive cohorts during the phase Ib portion to define the recommended phase II dose. Patients will continue gemcitabine, cisplatin, plus lenalidomide for up to 6 cycles, in the absence of disease progression or prohibitive toxicity. After completion of 6 cycles of therapy, patients who have achieved at least "stable disease" will proceed with "maintenance" lenalidomide given orally on days 1-21 of each 28-day cycle. Treatment will continue, in the absence of prohibitive toxicity, until the time of disease progression.
  Other Names: Revlimid

SUMMARY:
The primary objectives of this study are (Phase 1) to determine in subjects with unresectable or metastatic bladder cancer who have never had chemotherapy, the dose of lenalidomide that is well-tolerated when given in combination with gemcitabine plus cisplatin and (Phase 2) to study this recommended dose in subjects to evaluate progression-free survival at 1 year. The secondary objectives will be to determine the objective response rate to treatment, and the safety of combination therapy with gemcitabine, cisplatin and lenalidomide as well as to evaluate lenalidomide as maintenance treatment in subjects achieving objective response or stable disease.

DETAILED DESCRIPTION:
Urothelial carcinoma of the urinary bladder is the second most common genitourinary malignancy. Based on the results of a large randomized study comparing MVAC with gemcitabine plus cisplatin, the latter regimen became a treatment standard based on improved tolerability. While the tolerability of chemotherapy for patients with advanced urothelial carcinoma has improved, there have been no significant improvements in efficacy since the advent of MVAC in the 1980's and novel approaches are clearly needed.

The current study will explore the safety and activity of lenalidomide in combination with gemcitabine plus cisplatin as first line chemotherapy in subjects with metastatic urothelial carcinoma.

The primary objective of the phase Ib portion will be to determine the recommended phase II dose of the combination of gemcitabine, cisplatin, plus lenalidomide in patients with advanced/metastatic urothelial carcinoma. The primary objective of the phase II portion will be the progression-free survival at 1 year. The secondary objectives are to evaluate the activity (as determined by objective response rate); and to determine the safety (per the Common Terminology for Adverse Events version 4.0) of combination therapy with gemcitabine, cisplatin plus lenalidomide; to evaluate lenalidomide as maintenance treatment in patients achieving an objective response or stable disease following completion of 6 cycles of combination therapy and; to determine the impact of treatment on peripheral blood immune cell subsets and circulating tumor cells.

Patients will receive gemcitabine 1000 mg/m2 IV on days 1 + 8 and cisplatin 70 mg/m2 IV on day 1 of each 21 day cycle. Lenalidomide will be given orally on days 1-14 and the dose will be escalated in successive cohorts during the phase Ib portion to define the recommended phase II dose. Patients will continue gemcitabine, cisplatin, plus lenalidomide for up to 6 cycles, in the absence of disease progression or prohibitive toxicity. After completion of 6 cycles of therapy, patients who have achieved at least "stable disease" will proceed with "maintenance" lenalidomide given orally on days 1-21 of each 28-day cycle. Treatment will continue, in the absence of prohibitive toxicity, until the time of disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age > 18 years at the time of consent.
3. Karnofsky Performance Status of ≥ 70%.
4. Histological or cytological proof of transitional cell carcinoma of the urothelial tract. The primary site may include: urethra, bladder, ureters, and renal pelvis. Patients with mixed histologies may be enrolled provided that transitional cell carcinoma is the predominant histology.
5. Measurable disease according to RECIST or unresectable disease (cT4b).
6. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
7. Females of childbearing potential (FCBP)* must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control.
8. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).
9. Adequate organ function as determined by the following laboratory values:

   * Hemoglobin (Hgb) > 9 g/dL
   * Platelets > 100 x 1,000,000,000/L
   * Absolute neutrophil count (ANC) > 1.5 x 1,000,000,000/L
   * Calculated creatinine clearance of > 60 cc/min using the Cockcroft-Gault formula
   * Bilirubin < 1.5 x ULN
   * Aspartate aminotransferase (AST, SGOT) < 1.5 X ULN (< 5 X ULN if patient has hepatic metastases)

Exclusion Criteria:

1. Has had prior treatment with systemic chemotherapy for metastatic disease (prior intravesical therapy is permitted; prior neoadjuvant/adjuvant chemotherapy permitted if completed ≥ 1 year from study entry)
2. Has received prior lenalidomide.
3. Has had major surgery within 30 days of starting the study treatment
4. Has had any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
5. Has active CNS metastases. Subjects with neurological symptoms must undergo a head CT scan or brain MRI to exclude brain metastasis.
6. Has a history of a prior malignancy
7. Has received anticancer therapy, radiation, or any investigational agent within 30 days prior to being registered for protocol therapy.
8. Pregnant or breastfeeding.
9. Has a clinically significant infection as judged by the treating investigator.
10. Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Galsky, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - National Cancer Institute, Bethesda, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

REFERENCES:
- [Result] Agarwal N, Apolo AB, Tsao CK, Lee KM, Godbold JH, Soto R, Poole A, Gimpel-Tetra K, Lowe N, Oh WK, Galsky MD. Phase Ib/II trial of gemcitabine, cisplatin, and lenalidomide as first-line therapy in patients with metastatic urothelial carcinoma. Oncologist. 2014 Sep;19(9):915-6. doi: 10.1634/theoncologist.2014-0153. Epub 2014 Jul 22. PMID 25052451

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual at the Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah; the National Cancer Institute, Bethesda, Maryland;, and the Tisch Cancer Institute, Icahn School of Medicine at Mount Sinai, New York, NewYork over the course of 19 months.
Groups:
- Lenalidomide: lenalidomide in combination with gemcitabine and cisplatin (GCL) in patients with MUC
Period: Overall Study
Arm/Group | Lenalidomide
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 69 [44 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status:
  0 - Fully active, able to carry on all pre-disease performance without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. - Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  Participants
    0 | 0
    1 | 8
    2 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Lenalidomide
Description: MTD was determined by testing planned increasing doses up to 25 mg daily dose on days 1-14, starting at 10mg. MTD reflects the highest dose of drug that did not cause a Dose-Limiting Toxicity (DLT) in > 33% of participants. DLTs were defined as any lenalidomide-related Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE 4.0) Grade 3 or 4 adverse events
Time Frame: after 1 cycle (each cycle is 21 days)
Population: The dose of lenalidomide was not escalated beyond 10 mg because of cytopenias requiring repeated dose delays and reductions.
Measure: Number; unit: mg
Arm/Group | Lenalidomide
Number analyzed (Participants) | 9
mg | 10

2. Primary Outcome: Phase II: Progression-free Survival at 1 Year
Time Frame: 1 year
Population: Data not collected.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 0

3. Secondary Outcome: The Objective Response Rate to Treatment With Gemcitabine, Cisplatin, Plus Lenalidomide
Description: The objective response rate as determined by Response Evaluation Criteria in Solid Tumors (RECIST).
  Complete Response (CR) Disappearance of all target lesions for a period of at least one month.
  Partial Response (PR) At least a 30% decrease in the sum of the longest diameter of measures lesions (target lesions), taking as reference the baseline sum of the longest diameter.
  Stable Disease (NR/SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of the longest diameter since the treatment started.
  Progressive Disease (PD) A 20% or greater increase in the sum of the longest diameter of measured lesions (target lesions), taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: After 2 cycles (a cycle is 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 9
Participants
  CR | 1
  PR | 2
  SD | 3
  PD | 2
  not evaluable | 1

4. Secondary Outcome: Number of Grade >=3 Adverse Events
Description: Number of grade >=3 adverse events to assess the safety of combination therapy with gemcitabine, cisplatin plus lenalidomide as determined by the frequency and severity of adverse events as per the NCI Common Terminology for Adverse Events (CTCAE) version 4.0.
Time Frame: Day 1 and Day 8 of each treatment cycle; 21 days after the last dose of Lenalidomide
Measure: Number; unit: events
Arm/Group | Lenalidomide
Number analyzed (Participants) | 9
events
  Grade 3 | 28
  Grade 4 | 7

5. Secondary Outcome: Best Overall Response
Description: Best Overall Response to evaluate lenalidomide as maintenance treatment in patients achieving an objective response of either complete response or partial response following completion of 6 cycles of combination therapy.
  Complete Response (CR) - CR of target lesions and no new lesions Partial Response (PR) -PR of target lesions and no new lesions Stable Disease (SD) - SD of target lesions and no new lesions Progression Disease (PD) - any status of target lesions and new lesions
Time Frame: 168 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 9
Participants
  CR | 1
  PR | 2

6. Secondary Outcome: To Determine the Impact of Treatment on Peripheral Blood Immune Cell Subsets
Description: To determine the changes in cellular immunity with lenalidomide in peripheral blood mononuclear cells including Tregs, NK, NKT cells (Berg et al JCO 2010), sIl-2R, TNF alpha (Bartlett et al BJC 2004) and markers indicative of activation, i.e. CD107a. These analyses will only be done in the phase II portion of the protocol.
Time Frame: Day 1 of Cycle 0 and Day 1 of Cycle 2 (each Cycle is 21 days)
Population: Data not collected
Arm/Group | Lenalidomide
Number analyzed (Participants) | 0

7. Secondary Outcome: To Determine the Impact of Treatment on Circulating Tumor Cells
Description: Circulating epithelial tumor cells (CTC) will be investigated as an experimental endpoint using immunofluorescence techniques and CTC identification by positive expression of epithelial markers and a viability marker and negative expression of hematopoietic markers. These analyses will only be done in the phase II portion of the protocol.
Time Frame: Day 1 of Cycles 0, 1 and 2 (each Cycle is 21 days)
Population: Data not collected.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collected over the course of 19 months
Description: Listed are adverse events with grade 3 or higher
Groups:
- Lenalidomide for Cycle 1; Phase 2: lenalidomide in combination with gemcitabine and cisplatin (GCL) in patients with MUC
Arm/Group | Lenalidomide for Cycle 1 | Phase 2
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/9
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide for Cycle 1 (N=9) | Phase 2 (N=9)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide for Cycle 1 (N=9) | Phase 2 (N=9)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 2
ALP/ALT increase (General disorders) | 1 (1) | 1
Anemia (Blood and lymphatic system disorders) | 3 (3) | 1
Ascending Cholangitis (Hepatobiliary disorders) | 1 (1) | 0
Blurred Vision (Eye disorders) | 1 (1) | 0
Confusion (Nervous system disorders) | 1 (1) | 0
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0
Diarrhea (Gastrointestinal disorders) | 2 (2) | 6
Fatigue (General disorders) | 1 (1) | 4
Febrile neutropenia (Immune system disorders) | 1 (1) | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2
Hypomagnesium (Metabolism and nutrition disorders) | 1 (1) | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 2
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0
thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 5
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 3
Angular Chelitis (Gastrointestinal disorders) | 1 | 0
Anorexia (Gastrointestinal disorders) | 0 | 3
Bone pain (General disorders) | 0 | 1 — right midthigh and all pain
C. difficile infection (Gastrointestinal disorders) | 0 | 1
Cold (General disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Creatinine increased (Renal and urinary disorders) | 0 | 4
Dizziness (General disorders) | 0 | 4
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Edema (General disorders) | 0 | 4
Erythematous rash (Skin and subcutaneous tissue disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Flu-like symptoms (General disorders) | 0 | 1
Hand Tremors (General disorders) | 0 | 1
Hearing Loss (Ear and labyrinth disorders) | 0 | 2
Hematuria (Renal and urinary disorders) | 0 | 3
Hydrocephalus (Nervous system disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (General disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 2
Lightheadedness (General disorders) | 0 | 1
Loss of appetitie (General disorders) | 0 | 1
Lower back pain (General disorders) | 0 | 1
Mouth sores (Gastrointestinal disorders) | 0 | 2
Mucositis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 8
Neuropathy (Nervous system disorders) | 0 | 6
Oral Thrush (Gastrointestinal disorders) | 0 | 1
Pain extremities (General disorders) | 0 | 4
Phlebitis (Vascular disorders) | 0 | 2 — left lower leg
Pruritus (General disorders) | 0 | 1
Rhinorrhea (General disorders) | 0 | 1
Right-heel numbness (Nervous system disorders) | 0 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore Throat (General disorders) | 0 | 1
Syncope (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 2
Taste alteration (General disorders) | 0 | 2
Thromboembolism (Vascular disorders) | 0 | 4
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Urinary frequency (Renal and urinary disorders) | 0 | 1
Urinary hesitancy (Renal and urinary disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 8
Watering eye left (Eye disorders) | 0 | 1
Weakness (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The trial was terminated because the regimen was deemed poorly tolerated for chronic administration because of the need for repeated dose delays and reductions coupled with slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes